CLINICAL TRIAL: NCT06869525
Title: Study on the Efficacy and Mechanism of Acupuncture in the Acute Stage of Chronic Airway Diseases (Asthma and Chronic Obstructive Pulmonary Disease)
Brief Title: Study on Acupuncture Treatment of Chronic Airway Diseases(Asthma and Chronic Obstructive Pulmonary Disease)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCM for Chronic Airway Disease
Record Dates: First submitted 2025-02-18; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: COPD Exacerbation Acute; Asthma Acute
Keywords: COPD Exacerbation Acute; Asthma Acute; Acupuncture; Randomized Controlled Trial
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group for Asthma Acute/AECOPD (Experimental): Patients in the Asthma Acute/AECOPD experimental group were treated with Acupuncture
  Interventions: Behavioral: Acupuncture
- Sham Acupuncture group for Asthma Acute/AECOPD (Sham Comparator): Patients in the Asthma Acute/AECOPD experimental group were treated with Sham Acupuncture
  Interventions: Behavioral: Sham Acupuncture

INTERVENTIONS:
Behavioral: Acupuncture — Dingchuan, Shanzhong, Tiantu, Feishu, Kongji, after obtaining qi, connect the electric needle (continuous wave, The frequency was 2Hz, the current intensity was 1~5mA, and the current intensity was gradually increased according to patient tolerance), and the treatment was 30min.
  Arms: Acupuncture group for Asthma Acute/AECOPD
Behavioral: Sham Acupuncture — Dingchuan, Shanzhong, Tiantu, Feishu, hole the most points open 5~10mm, shallow piercing through the skin, connected with the electric needle but no electricity, treatment 30min.
  Arms: Sham Acupuncture group for Asthma Acute/AECOPD

SUMMARY:
For patients in the acute phase of chronic airway diseases, on the basis of guideline-directed treatment, the experimental group was given acupuncture treatment, while the control group was given sham acupuncture treatment. The treatment lasted for one week, followed by a 13-week follow-up. For asthma and COPD, PEF and CAT were respectively used as the primary outcome measures to evaluate the clinical efficacy and safety of acupuncture. Based on the improvement of the primary outcome measures, the advantageous population was identified. The mechanism by which acupuncture reduces airway mucus hypersecretion was preliminarily explained.

DETAILED DESCRIPTION:
This study was a multicenter, randomized, double-blind, controlled trial. A total of 336 patients with acute exacerbation of chronic obstructive pulmonary disease (COPD) and 240 patients with acute attack of asthma were included. On the basis of guideline-directed treatment, the experimental group received acupuncture treatment, while the control group was given sham acupuncture treatment. For patients with AECOPD, the acupoints selected were Zhongfu, Dingchuan, Tiantu, Fenglong, and Feishu. For patients with acute attack of asthma, the acupoints selected were Dingchuan, Zhongfu, Tiantu, Feishu, and Kongzui. The acupoints were connected to electroacupuncture and treated for 30 minutes. The control group received sham acupuncture treatment. The acupoints were located 5 to 10 mm away from the actual acupoints, and the needles were inserted superficially through the skin. The acupoints were connected to electroacupuncture but without electricity. The treatment lasted for 30 minutes, once a day, for one week. Follow-up was conducted for 13 weeks. For COPD, the COPD Assessment Test (CAT) was the primary outcome measure, and the secondary outcome measures included the mMRC scale, assessment of airway mucus hypersecretion, CT assessment of airway mucus, basic vital signs, clinical symptom scores, use of control medications and antibiotics, acute exacerbation status, hospitalization time, tracheal intubation rate, and arterial blood gas. For asthma, the peak expiratory flow (PEF) was the primary outcome measure, and the secondary outcome measures included the Asthma Control Test (ACT), Asthma Control Questionnaire (ACQ), Asthma Quality of Life Questionnaire (AQLQ), assessment of airway mucus hypersecretion, CT assessment of airway mucus, basic vital signs, clinical symptom scores, use of control medications and antibiotics, acute attack status, hospitalization time, and fractional exhaled nitric oxide (FeNO). The clinical efficacy and safety of acupuncture were evaluated. The population with advantages was identified based on the improvement of the primary outcome measures. The mechanism of acupuncture in reducing airway mucus hypersecretion was preliminarily explained.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for acute attack of asthma/AECOPD;
* Age range from18 years to 80 years(asthma) and 40 yesrs to 80 years(COPD);
* The investigators agreed to participate in this clinical study by voluntarily signing an informed consent form.

Exclusion Criteria:

* Patients with combined pulmonary abscess, pulmonary interstitial fibrosis, active pulmonary tuberculosis, bronchiectasis and other pulmonary diseases;
* Patients with severe cardiovascular and cerebrovascular diseases (such as malignant arrhythmia, unstable angina pectoris, acute myocardial infarction, grade 3 or above cardiac function, stroke, cerebral hemorrhage, etc.);
* Patients with severe liver diseases (such as liver cirrhosis, portal hypertension and bleeding caused by esophageal and gastric fundus varices) and severe kidney diseases (such as dialysis, kidney transplantation, etc.);
* Patients with impaired consciousness or various mental disorders who are unable to communicate normally;
* Pregnant and lactating women;
* Those who are currently participating in other clinical trials within 1 month before enrollment;
* Patients with contraindications to acupuncture (such as severe allergic or infectious skin diseases);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Astham part: PEF | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  Record the peak expiratory flow rate(PEF) for each patient, and evaluate the impact of acupuncture on improving the peak expiratory flow (PEF) of asthma patients.
COPD part：CTA | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  Record the COPD Assessment Test (CAT) for each patient, and evaluate the impact of acupuncture on improving the clinical symptoms of patients with AECOPD.

SECONDARY OUTCOMES:
Astham part: the Asthma Control Test (ACT) | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  ACT includes five questions. Every question will be assessed using a 5-point scale with scores ranging from 5 to 25. The higher the score, the better the symptom control.25 is considered complete control level, 20 ~ 24 is considered good control level, and <20 is considered non-control level.
Asthma part：Asthma Control Questionnaire(ACQ) | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  The content of ACQ involves the following aspects: asthma-related, symptoms, the use of first-aid drugs, the impact on daily life and lung function test results.The higher the score, the worse the state.
Asthma part：Asthma Quality of Life Questionnaire(AQLQ) | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  The asthma quality of life scale (5-point scale-RRB- consists of 35 items, including activity limitation (1-12) , asthma symptoms (13-20) , psychological status (22-26) , response to stimuli (27-31) , concern for one's own health (32-35) . On a 5-point scale, 1 is the worst and 5 is the best.
Asthma part：The cough and expectoration assessment questionnaire (CASA-Q) | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  Each indicator of the patient is scored from 1 to 5 based on the severity. After reverse scoring, the lower the score, the more severe the airway mucus hypersecretion and the poorer the therapeutic effect.
Asthma part：Evaluation of Airway Mucus Hypersecretion | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  The assessment includes: the difficulty of expectoration score, the sputum character score, and the sputum viscosity grading. They represent the nature of the sputum and the difficulty of coughing, ranging from 0 to 3 points. The higher the score, the more mucus secretion in the airway and the more severe the symptoms.
Asthma part：Evaluation of Airway Mucus by CT Imaging | Before treatment, and day 7
  Airway mucus CT assessment evaluates the distribution characteristics of airway mucus through the imaging features of thin-layer CT.
Asthma part：Clinical symptom score | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  Including wheezing, coughing, expectoration, chest tightness and wheezing sounds.A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
Asthma part：Acute attack status | Follow-up at the 4th and 13th weeks
  Including the number and severity of acute attacks, the re-admission rate after acute attacks, and the interval between the first acute attack and the subsequent ones.
Asthma part：Hospitalization time | At 4 weeks of follow-up
  The time required from the point of enrollment to the attainment of the discharge criteria
Asthma part：Fractional exhaled nitric oxide (FeNO) | Before treatment, and day 7
  FeNO is measured by a FeNO detector. It is used to determine the concentration of nitric oxide in exhaled breath of the human body. As a biomarker of airway inflammation, its normal range is less than 25ppb (adults) .
COPD part：clinical symptoms and signs questionnaire | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  Assessment will be performed by clinical symptoms and signs questionnaire. The clinical symptoms to be evaluated in this study include cough, phlegm, chest tightness, gasp,shortness of breath, feeble and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
COPD part：mMRC | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "4" means severe dyspnea perception.
COPD part：The cough and expectoration assessment questionnaire (CASA-Q) | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  Each indicator of the patient is scored from 1 to 5 based on the severity. After reverse scoring, the lower the score, the more severe the airway mucus hypersecretion and the poorer the therapeutic effect.
COPD part：Evaluation of Airway Mucus Hypersecretion | Before treatment, at 4 and 7 days of treatment, and at 4 and 13 weeks of follow-up
  The assessment includes: the difficulty of expectoration score, the sputum character score, and the sputum viscosity grading. They represent the nature of the sputum and the difficulty of coughing, ranging from 0 to 3 points. The higher the score, the more mucus secretion in the airway and the more severe the symptoms.
COPD part：Evaluation of Airway Mucus by CT Imaging | Before treatment, and day 7
  Airway mucus CT assessment evaluates the distribution characteristics of airway mucus through the imaging features of thin-layer CT.
COPD part：Acute attack status | Follow-up at the 4th and 13th weeks
  The number of acute attacks
COPD part：Hospitalization time | At 4 weeks of follow-up
  The time required from the point of enrollment to the attainment of the discharge criteria
COPD part：Tracheal intubation rate | At 4 weeks of follow-up
  The proportion of patients with tracheal intubation during the treatment period;
COPD part: Arterial blood gas | Before treatment, and day 7
  The arterial blood PaO2, PaCO2 of the two groups of subjects were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Suyun Li, Professor, Study Chair — First Affiliated Hospital of Henan University of Traditional Chinese Medicine